CLINICAL TRIAL: NCT01039259
Title: The Impact of Material on Microbiota in Association With Tongue and Lip Piercing
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Collaborators: Austrian Society of Periodontology (Other)
Responsible Party: Ines Kapferer, Dr., Innsbruck Medical University
Other Study IDs: AN3223 265/4.7
Record Dates: First submitted 2009-12-23; First posted 2009-12-24 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-01

CONDITIONS: Bacteremia
Keywords: adolescent; body piercing/adverse effects; tongue piercing; tongue/microbiology
MeSH Terms: conditions — Bacteremia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- subjects with lip piercing
  Interventions: Device: piercings of four different materials
- subjects with tongue piercing
  Interventions: Device: piercings of four different materials

INTERVENTIONS:
Device: piercings of four different materials — randomly assigned sterile piercings are inserted for two weeks
  Other Names: piercing materials:; steel, titanium, polypropylene, polytetrafluoroethylene

SUMMARY:
Biofilms on oral piercings may serve as a bacterial reservoir and lead to systemic bacteraemia or local transmission of periopathogenic microbiota.

The investigators hypothesize that there are microbiological differences in bacterial samples collected from tongue /or lip piercings made of different materials. The investigators also hypothesize that the piercings carry the same characteristic bacteria as found in the piercing channels and that independently the biofilm on the tongue/adjacent teeth is similar to the other study locations.

85 subjects with tongue and 85 subjects with lip piercing will participate. Periodontal clinical parameters, traumata of hard tissues, and characteristics of the stud are evaluated. Sterile piercings of four different materials will be randomly allocated to the study subjects. After two weeks, microbiologic samples are collected and are processed by checkerboard DNA-DNA hybridization methods.

ELIGIBILITY:
Inclusion Criteria:

* lip/tongue piercing for at least six month in situ

Exclusion Criteria:

* pregnancy and lactating women
* medication with known effects on gingival tissues
* antibiotic medication in the last six months or need for antibiotic prophylaxis
* chlorhexidine use in the last six months
* non-plaque induced gingival disease
* prior diagnosis of periodontitis

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 85 subjects with lip piercing 85 subjects with tongue piercing
Sampling Method: Probability Sample
Enrollment: 170
Dates: Start 2008-08; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
microbiologic findings of piercing samples | 2 weeks

SECONDARY OUTCOMES:
microbiologic findings in piercing channels, microbiologic findings on the tongue/adjacent teeth | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ines Kapferer, Dr., Principal Investigator — Innsbruck Medical University
Locations (1):
- Innsbruck Medical University, Innsbruck, Austria